CLINICAL TRIAL: NCT07380217
Title: Use of mechaNical Left ventricuLar unlOADing in Complex Higher-risk Indicated Procedures
Acronym: UNLOAD-CHIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Pulsecath BV. (Unknown)
Responsible Party: Principal Investigator, Alexander Nap, Principal investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL83524.018.23; NL-OMON53381 (Other: International Clinical Trials Registry Platform)
Record Dates: First submitted 2026-01-08; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: High-risk PCI; Coronary Artery Disease Risk High
Keywords: High-risk PCI; CHIP; Mechanical Circulatory Support; Pulsecath iVAC2L; Pulsecath; iVAC2L

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard-of-Care (without MCS) (No Intervention): Patients will undergo high-risk PCI without upfront use of MCS
- Pulsecath iVAC2L (with MCS) (Experimental): Patients will undergo high-risk PCI with upfront use of the Pulsecath iVAC2L (MCS)
  Interventions: Device: Mechanical circulatory support with the Pulsecath iVAC2L device

INTERVENTIONS:
Device: Mechanical circulatory support with the Pulsecath iVAC2L device — The Pulsecath iVAC2L is a pulsatile pump, placed in the left ventricle, that ejects blood into the ascending aorta at a flow up to 2L/min. Theoretically, pulsatility maintains the physiological vascular responses and endothelial function at the level of the -systemic and -micro circulation and might offer benefit when compared to continues flow devices such as Impella. In contrast, IABP (which also offers pulsatile support), lacks the possibility of active unloading. Therefore, the combination of those features in the PulseCath iVAC2L is unique.
  Arms: Pulsecath iVAC2L (with MCS)

SUMMARY:
If there is a narrowing or blockage in the coronary arteries of the heart, the cardiologist may choose to treat this blockage. This is called percutaneous coronary intervention (PCI), which involves both balloon angioplasty and the placement of a stent. PCI is a commonly performed and safe procedure. However, in your case, the procedure is more complicated than usual due to the location and nature of the narrowing, the required technique for the intervention, and the fact that your heart function is reduced. As a result, your PCI will carry a higher risk than usual.

During the procedure, balloons are inflated to clear the blockage, and a stent is placed to keep the artery open. This temporarily reduces or even stops the blood and oxygen supply to a large portion of the heart. This moment presents a higher risk for complications, such as low blood pressure or cardiac arrest. As a result, the heart may not pump blood effectively throughout the body, which can lead to oxygen deprivation in other organs.

To help the heart in this situation, it is possible to insert a mechanical heart pump during the procedure. This form of support is introduced via an artery in the groin into your left ventricle. The pump helps the heart function and may improve the circulation to the body's organs. On the other hand, the placement of the pump increases the chance of complications. Therefore, there are both potential benefits and risks. It is currently unclear whether PCI with the temporary pump can be performed more safely than without it.

This study aims to investigate whether mechanical circulatory support, specifically with the Pulsecath iVAC2L, leads to improved outcomes for patients undergoing high-risk PCI.

DETAILED DESCRIPTION:
During the last three to four decades percutaneous coronary intervention (PCI) tools and techniques have improved immensely. Currently, PCI is the most widely used approach for myocardial revascularization. In general, elective PCI is considered a safe and relatively low-risk procedure.

However, patients with left main or complex coronary lesions or impaired left ventricular function remain at high risk for peri-procedural and post-procedural hemodynamic instability and death.

Mechanical circulatory support (MCS) devices, such as intra-aortic balloon pump (IABP) and Impella (Impella 2.5 and CP), have emerged as potential tools to avoid hemodynamic instability during these CHIP coronary interventions. These devices have shown to improve hemodynamics / cardiac output during complex PCI procedures, although the benefit of mechanical circulatory support in CHIP PCI remains debated and no clear benefit on patient outcomes has been shown. A recent large scale analysis favoured Impella as opposed to IABP. The use of these devices, especially Impella, is associated with increased risk for complications such as bleeding. The use of MCS for optimizing peri-procedural hemodynamic support needs to be balanced out against the potential risk for MCS related complications.

Recently the PulseCath iVAC 2L was introduced. This is a pulsatile pump, placed in the left ventricle, that ejects blood into the ascending aorta at a flow up to 2L/min. Theoretically, pulsatility maintains the physiological vascular responses and endothelial function at the level of the -systemic and -micro circulation and might offer benefit when compared to continues flow devices such as Impella. In contrast, IABP (which also offers pulsatile support), lacks the possibility of active unloading. Therefore, the combination of those features in the PulseCath iVAC2L is unique.

Recent studies performed with the PulseCath iVAC2L in the setting of CHIP PCI demonstrated hemodynamic advantages with afterload reduction, increased stroke volume and higher cardiac output. Also, the device was deemed safe in terms of complications. Samol et al. showed in a prospective cohort study that the use of IVAC2L was non-inferior to Impella in terms of feasibility and safety, even if complications occur. Other advantages of the IVAC2L are its relatively simple use and lower costs when compared to other mechanical circulatory support devices such as the Impella family. Considering that the IVAC2L is powered by an IABP console, the possibility of widespread use adds an even greater advantage.

So far, MCS facilitated CHIP has not been proven beneficial compared to a conservative (non-supported) high-risk procedure. Although high-risk criteria parameters such as coronary anatomy (location and complexity), co-morbid conditions, and concomitant cardiac disease (structural or valvular disease, left ventricular dysfunction) are well known, no intrinsic value of each of these components is determined. The recent PULSE trial shed some light on this gap of knowledge by showing possible additional hemodynamic benefit for patients with mitral regurgitation, who presented with an acute coronary syndrome (ACS) and who had higher cardiac filling pressures at baseline. Therefore, MCS-facilitated high-risk PCI might be beneficial if used in ACS patients or patients with (left-sided) congestion (stabilized acutely decompensated heart failure) with low hemodynamic tolerance. However, due to the low number of patients enrolled and non-randomized nature of this study, conclusions should be drawn with caution. To this day, no randomized controlled trials have been executed with the PulseCath iVAC2L in this subset of CHIP patients who are thought to benefit from an MCS-facilitated PCI. Its place in the setting of CHIP PCI remains to be elucidated.

Research hypothesis:

Prophylactic percutaneous mechanical left ventricular unloading by insertion of the PulseCath iVAC2L during complex coronary stenting (complex left main disease or equivalent or last remaining vessel) at risk for prolonged procedural ischemia in patients with severely reduced LV function is superior to a mechanical unassisted PCI procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years AND
* Multidisciplinary heart team consensus for high risk PCI +/- MCS AND
* Hemodynamically stable (SCAI A-B) AND
* LVEF <30% OR LVEF <35% with moderate MR OR LVEF <40% with severe MR AND
* Complex left main disease (calcium modifying techniques deemed necessary OR 2-stent techniques, left dominant system) OR equivalent (ostial LAD and RCX) OR last remaining vessel (native).

Exclusion Criteria:

* Contraindications for Pulsecath IVAC2L:

  1. severe aortic regurgitation
  2. known presence of an LV thrombus (contrast echo/MRI)
  3. Mechanical aorta valve prosthesis
  4. severe aortic valve stenosis
  5. peripheral arterial disease that would preclude placement of the PulseCath iVAC2L device
* Cardiogenic shock defined as either SCAI CSWG stage C-E
* Patient is intubated and mechanically ventilated
* Stroke <3 months
* Major bleeding event <3 months
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombo-cytopenia), any recent GU or GI bleed, or will refuse blood transfusions.Renal replacement therapy
* Pregnancy, or suspected thereof.
* BMI > 35
* Other medical, social, or psychological problems that, in the opinion of the Investigator, compromises the subject's ability to give written informed consent and/or to comply with study procedures.
* Subject belongs to a vulnerable population (defined as individuals with mental disability, persons in nursing homes, impoverished persons, homeless persons, nomads, refugees and those permanently incapable of giving informed consent; vulnerable populations also may include members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the Sponsor, members of the armed forces and persons kept in detention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint: - All-cause death - Cardiogenic shock (SCAI stage C-E) - (Need for) renal replacement therapy - (Need for) mechanical ventilation - Ventricular arrhythmias leading to loss of cardiac output requiring CPR | 30 days

SECONDARY OUTCOMES:
PCWP (Δ max) | Periprocedural
LVEDP (Δ max) | Periprocedural
CO / CI / CPO (Δ max) | Periprocedural
SvO2 (Δ max) | Periprocedural
Drop in arterial pressure (MAP <60 OR SBP <90) for >10 minutes | Periprocedural
Protected procedural success of Pulsecath iVAC2L | Periprocedural
  Proper placement and circulatory support of the device. Moreover, the device should be successfully weaned on the cardiac catheterization laboratory and maximally within 1 hour post CHIP procedure.
Procedural success of Pulsecath iVAC2L | <6 hours post-PCI
  Proper placement and circulatory support of the device. Moreover, the device should be successfully weaned <6h post-procedural.
Rescue pVAD implantation | From index PCI through hospital discharge (up to 30 days)
Highest Vasoactive Inotropic Score | From index PCI through hospital discharge (up to 30 days)
Length of hospital stay | From index PCI through hospital discharge (up to 30 days)
Cardiovascular death | 30 days
Major adverse cardiovascular cerebral events (MACCE) | 30-days
Stroke | 30-days
PCI related myocardial infarction | 48 hours
Myocardial infarction >48 hours post-PCI | 30-days
Re-hospitalization or urgent hospital visit for heart failure | 30 days

OTHER OUTCOMES:
Major vascular events | 30 days
  Safety endpoint
Limb ischemia | 30 days
  Safety endpoint
Bleeding events (BARC 3 and 5) | 30 days
  Safety endpoint
Aortic valve injury | 30 days
  Safety endpoint

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Amsterdam University Medical Center, Amsterdam
  - Zuyderland, Geleen
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Haaglanden Medical Center, The Hague
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
The publication rights in regard to the main results of the trial, i.e., regarding the primary and secondary objectives, belong to the sponsor. No individual investigator may publish on the results of this trial, or their own patients, without prior approval from the sponsor.
Supporting Information: Study Protocol

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: First approved protocol (version 4) (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT07380217/Prot_SAP_000.pdf
  • Study Protocol: Amendment (version 5) (2024-10-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT07380217/Prot_001.pdf